CLINICAL TRIAL: NCT00000301
Title: Rapid Evaluation of Cocaine Pharmacotherapies (Amantadine)
Brief Title: Rapid Evaluation of Amantadine for Treatment of Cocaine Abuse/Dependence - 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09260-4; P50DA009260 (NIH); P50-09260-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Cocaine-Related Disorders
Keywords: Amantadine; Cocaine; Pharmacotherapy; Outpatient
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Amantadine

INTERVENTIONS:
Drug: Amantadine

SUMMARY:
The purpose of this study is to empirically test a series of medications to: 1) determine each medication's efficacy in treatment of cocaine abuse/dependence; 2) find most effective dose range for each medication. In this study, amantadine is tested."

DETAILED DESCRIPTION:
16-week participation plus a 2 weekk lead-in period. Participants are assigned randomly to placebo or amantadine. Participants attend group meeting 3 times/week

ELIGIBILITY:
Inclusion Criteria:

M/F, ages 18-65. cocaine dependence according to DMS-IV criteria. Self-reported use within the last 30 days. Agreeable to conditions of the study and signed informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy, history of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative-hypnotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1996-03; Primary Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
Retention
Cocaine use
Cocaine craving
Psychosocial progress

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Shoptaw S, Kintaudi PC, Charuvastra C, Ling W. A screening trial of amantadine as a medication for cocaine dependence. Drug Alcohol Depend. 2002 May 1;66(3):217-24. doi: 10.1016/s0376-8716(01)00205-8. PMID 12062456